CLINICAL TRIAL: NCT05384717
Title: Do Fidget Instruments Enhance Attentional Control and Comprehension in 6-13 Year-olds With Attention Deficit Hyperactivity Disorder (ADHD)?
Brief Title: Examining the Impacts of Fidget Technology on Attention in Children With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: 3-C Family Services (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22-0531
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-05

CONDITIONS: ADHD
Keywords: Fidget technology; ADHD; Children; Developmental Psychology
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fidget group (Experimental): Participants in the experimental fidget group select a fidget from 4 options: fidget spinner, stress ball, pop-it, or fidget cube
  Interventions: Other: Fidget Device
- Control group (Placebo Comparator): No fidget choice provided
  Interventions: Other: Control group

INTERVENTIONS:
Other: Fidget Device — Fidget spinner, stress ball, pop-it, or fidget cube
  Arms: Fidget group
Other: Control group — No intervention
  Arms: Control group

SUMMARY:
Purpose: The purpose of this study is to investigate the usage of fidget technology and its effects on attention, working memory, and comprehension in children ages 6-13 with Attention Deficit Hyperactivity Disorder (ADHD). This study aims to examine the implications of fidget usage 2 different measures of attention; attentional control (working memory domain) and comprehension (recall, encoding, and recognition).

Participants: 6-13 year-old clients at 3-C Family Services, a private mental health clinic in Cary, NC, with a diagnosis of ADHD (Inattentive, Hyperactive, or combined types). Exclusion criteria: participants with an Intelligence Quotient (IQ) below 70 as estimated by referring 3-C clinical staff, or any history of psychosis.

Procedures (methods): This research will use a demographic and background collecting survey to gather relevant data about each participant. Parents will be asked to fill out a baseline ADHD Rating Scale-IV: Home Version (ADHD-RS), to account for their child's symptoms of ADHD over the past 6 months. Participants will be randomly assigned to one of 2 conditions, an experimental group where participants select a fidget, and a control group where participants are not provided a fidget. Fidget options will include a fidget spinner, pop-it, stress ball, and fidget cube as not all children would benefit from the same type of fidget equally. Participants in the experimental group will then be allowed to practice with and familiarize themselves with the fidget for 1 minute to decrease the attentional drain that the fidget may pose in its initial state.

After random assignment to either control or experimental group, participants in each group will then complete the same 2-back version of the N-back Attention Control Task (cognitivefun.net), and a video comprehension multiple choice test. After 3 minutes N-back scores will be recorded including visual correct ratio and visual response time scores. The video comprehension item is adapted from Lee and List, 2019. The video is a Ted Talk titled "The Survival of the Sea Turtle" ( https://www.youtube.com/watch?v=t-KmQ6pGxg4). Items in the multiple choice test will be aggregated to a score of percent correctness for each participant. Participants may request to have questions read to them by the research assistant present.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADHD

Exclusion Criteria:

* Psychosis
* IQ under 70

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-09-24 (Actual)

PRIMARY OUTCOMES:
N-back Visual correct ratio | Day 1 (Up to 30 minutes)
  The N-Back task is a measure of working memory. Participants are presented a sequence of stimuli and must decide if the current stimulus is the same as the one presented two trials ago. Max value= 1, min value =0, higher scores are closer to 1
N-back visual response time | Day 1 (Up to 30 minutes)
  The N-Back task is a measure of working memory. Participants are presented a sequence of stimuli and must decide if the current stimulus is the same as the one presented two trials ago. The lower the score the better (indicates less time to decide on n-back). For response time measure there is no minimum or maximum.
Number of correct multiple choice responses out of 10 | Day 1 (Up to 30 minutes)
  Participants answer 10 multiple choice questions to assess comprehension of Ted Talk video. Multiple choice questions adapted from Lee & List, 2019. Max value= 10, min value = 0. Best possible score = 10, higher scores are better.

SECONDARY OUTCOMES:
ADHD-RS Home Version Score | Day 1 (Up to 30 minutes)
  Parents complete a 18 question assessment of child's ADHD symptoms over the past 6 months. Max score= 54, Min score= 0. Higher score indicates more ADHD symptoms.
Parent-reported type of ADHD | Day 1 (Up to 30 minutes)
  Parents indicate the type of ADHD their child presents with. Categorical variable: Inattentive, Hyperactive, or Combined
Type of fidget selected | Day 1 (Up to 30 minutes)
  4 choices of fidget are available to each participant in the experimental group. Categorical variable- fidget spinner, stress ball, pop-it, or fidget cube

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer R Persia, Principal Investigator — University of North Carolina, Chapel Hill; Steven G Buzinski, Study Chair — University of North Carolina, Chapel Hill; Lori A Schweickert, Study Director — 3-C Family Services
Locations (1):
- 3-C Family Services, Cary, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: beginning 9 to 36 months following publication
Access Criteria: Researcher has approved from an IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Result] Lee, Hye Yeon & List, Alexandra. (2019). Processing of texts and videos: A strategy-focused analysis. Journal of Computer Assisted Learning. 35. 10.1111/jcal.12328